CLINICAL TRIAL: NCT05340088
Title: Optimal Passive Dilation Time in Retrograde Intrarenal Surgery
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yildiz, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: DJRIRS2022
Record Dates: First submitted 2022-03-30; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Stone, Kidney; Urolithiasis
MeSH Terms: conditions — Kidney Calculi; Urolithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who underwent RIRC for 2-4 weeks after DJ stent placement for passive dilatation: Patients who underwent RIRC for 2-4 weeks after DJ stent placement for passive dilatation
  Interventions: Procedure: Retrograde intrarenal surgery after DJ stent placement
- Patients who underwent RIRC for 4-6 weeks after DJ stent placement for passive dilatation: Patients who underwent RIRC for 4-6 weeks after DJ stent placement for passive dilatation
  Interventions: Procedure: Retrograde intrarenal surgery after DJ stent placement

INTERVENTIONS:
Procedure: Retrograde intrarenal surgery after DJ stent placement — Patients who underwent RIRC for 2-4 weeks after DJ stent placement for passive dilatation

SUMMARY:
Retrograde intrarenal surgery (RIRC) is used as standard treatment for stones less than 2 cm. In some cases, the ureteral access sheath cannot be placed due to ureteral stricture. In this case, a double j stent (DJ) is placed to passively dilate the ureter, and the RIRC is postponed for post-dilatation. The aim of the study is to determine the optimal time for RIRC operation in cases where a double j stent was placed for passive dilatation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a DJ stent for passive dilatation and subsequent RIRC

Exclusion Criteria:

* Urinary tract infection, patients with ureteral compression and a history of pelvic radiotherapy, urinary system tumor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a DJ stent for passive dilatation and subsequent RIRC
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
BMI in kg/m^2 | 3 Months
  BMI in kg/m^2the kidney, operation time(minute)
serum creatinine mg/dl | 3 Months
  serum creatinine mg/dl

SECONDARY OUTCOMES:
mm size of the stone | 3 Months
  mm size of the stone
localization of the stone in the kidney, | 3 Months
  localization of the stone in the kidney,

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bai PD, Wang T, Huang HC, Wu Z, Wang XG, Qin JX, Wang HQ, Chen B, Hu MB, Xing JC. Effect of Preoperative Double-J Ureteral Stenting before Flexible Ureterorenoscopy on Stone-free Rates and Complications. Curr Med Sci. 2021 Feb;41(1):140-144. doi: 10.1007/s11596-021-2328-z. Epub 2021 Feb 13. PMID 33582918
- [Background] Yuk HD, Park J, Cho SY, Sung LH, Jeong CW. The effect of preoperative ureteral stenting in retrograde Intrarenal surgery: a multicenter, propensity score-matched study. BMC Urol. 2020 Sep 14;20(1):147. doi: 10.1186/s12894-020-00715-1. PMID 32928162